CLINICAL TRIAL: NCT03188458
Title: Immunogenicity of a Single Dose of GSK Biologicals' Diphtheria, Tetanus and Acellular Pertussis (dTpa) Booster Vaccine (Boostrix™ [263855]) in Infants Prior to Primary Pertussis Vaccination, When Administered to Pregnant Women as Per Routine Practice in Bogota, Colombia
Brief Title: Immunogenicity of a Single Dose of GSK Biologicals' Boostrix™ in Infants Prior to Primary Pertussis Vaccination, When Administered to Pregnant Women as Per Routine Practice in Bogota, Colombia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: As similar local evidence recently available, present study will not add new information; no ethical justification exists to continue study procedures.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201522
Record Dates: First submitted 2017-05-19; First posted 2017-06-15 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Diphtheria-Tetanus-Acellular Pertussis
Keywords: Infants; Cord blood sample; Acellular pertussis; Boostrix; Colombia; Pregnant women
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Second and third trimester Group (Other): This study group will include infants whose mothers have received Boostrix during the second (21-27 weeks) and third trimester (above 28 weeks) of their pregnancy, as per routine practice.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood samples will be collected from infants prior to their first routine primary pertussis vaccination (At Visit 2 [approximately 4-8 weeks of age]).

SUMMARY:
The purpose of the study is to support the recommendation of vaccination of all pregnant women in Colombia with Diptheria, tetanus and pertussis (dTpa) by studying the transfer of pertussis specific IgG antibodies from mother to the child.

DETAILED DESCRIPTION:
This study will assess the immunogenicity in infants (at birth and just prior to primary pertussis vaccination [i.e. diphtheria, tetanus and pertussis [DTP] vaccination] administered at 8 weeks of age), of a single Boostrix booster dose administered to their mothers during the second or third trimester as per routine practice in Bogota, Colombia.

ELIGIBILITY:
Inclusion Criteria:

Criteria applicable at screening (before the birth of the infant):

* Male or female infants whose mothers have received Boostrix during their current pregnancy, as per routine practice.
* Infant whose parents, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from both parents of the infant.

Criteria applicable at enrolment (after the birth of the infant):

* Confirmation of written informed consent obtained from both parents of the infant at the time of screening.
* Infant whose parents, in the opinion of the investigator, can and will comply with the requirements of the protocol.

Exclusion Criteria:

Criteria applicable at screening (before the birth of the infant):

* Infants whose parents are below the legal consenting age of the country.
* Infant's whose mother has multiple pregnancies.
* Infant's whose mother has any confirmed or suspected immunosuppressive or immunodeficient condition (including positive infection with human immunodeficiency virus [HIV]), based on medical history, physical examination or positive test result.
* Infant's whose mother is concurrently participating in another clinical study, at any time during the study period, in which the infant's mother has been or will be exposed to an investigational or a non-investigational vaccine/product.

Criteria applicable at enrolment (after the birth of the infant):

* Child in care.
* In case of multiple births.
* Infants with any confirmed or suspected immunosuppressive or immunodeficient condition , based on medical history, physical examination or positive test result.
* Infants who are concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Number of seropositive subjects for anti-pertussis toxin (PT), anti-filamentous haemagglutinin (FHA) and anti-pertactin (PRN). | For cord blood sample - Visit 1 (Day 0). For blood samples collected from infants prior to their first routine primary pertussis vaccination - Visit 2 (at approximately 4-8 weeks of age of subjects).
  Seropositivity status was defined as anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 EL.U/mL.

SECONDARY OUTCOMES:
Number of seropositive subjects for anti-PT, anti-FHA and anti-PRN. | At birth (Day 0) and before primary vaccination (between Day 28 and Day 56).
  Seropositivity status was defined as anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 EL.U/mL.
Anti-PT, anti-FHA and anti-PRN antibody concentrations. | At birth (Day 0) and before primary vaccination (between Day 28 and Day 56).
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off of 5 EL.U/mL.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.